CLINICAL TRIAL: NCT03760718
Title: Chloroprocaine Lavage to Improve Outcomes Related to Operative Cesarean Delivery
Acronym: CLOR-PRO
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Brandon M Togioka, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19021
Record Dates: First submitted 2018-11-09; First posted 2018-11-30 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Cesarean Section
Keywords: chloroprocaine; cesarean delivery; lavage
MeSH Terms: interventions — chloroprocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Preservative free Chloroprocaine Group 1 (Active Comparator): 40 ml of preservative-free 1% chloroprocaine
  Interventions: Drug: Preservative free 1% Chloroprocaine
- Preservative free Chloroprocaine Group 2 (Active Comparator): 40 ml of preservative-free 2% chloroprocaine
  Interventions: Drug: Preservative free 2% Chloroprocaine
- Preservative free Chloroprocaine Group 3 (Active Comparator): 40 ml of preservative-free 3% chloroprocaine
  Interventions: Drug: Preservative free 3% Chloroprocaine

INTERVENTIONS:
Drug: Preservative free 1% Chloroprocaine — 40 ml of preservative-free 1% chloroprocaine is planned for administration into the peritoneal cavity after delivery of the baby.
  Other Names: Nesacaine
  Arms: Preservative free Chloroprocaine Group 1
Drug: Preservative free 2% Chloroprocaine — 40 ml of preservative-free 2% chloroprocaine is planned for administration into the peritoneal cavity after delivery of the baby.
  Other Names: Nesacaine
  Arms: Preservative free Chloroprocaine Group 2
Drug: Preservative free 3% Chloroprocaine — 40 ml of preservative-free 3% chloroprocaine is planned for administration into the peritoneal cavity after delivery of the baby.
  Other Names: Nesacaine
  Arms: Preservative free Chloroprocaine Group 3

SUMMARY:
The long term objective is to show that intraperitoneal chloroprocaine can be used an alternative option to avoid general anesthesia during cesarean delivery, to alleviate mother's discomfort from surgical pain, reduce complications, and improve the birth experience. The objectives in this study are to determine the amount of chloroprocaine that is absorbed into the blood in order to create a plasma concentration time profile and to determine the incidence of side effects to help guide selection of an appropriate concentration for future study.

DETAILED DESCRIPTION:
Compared to general anesthesia, neuraxial anesthesia (spinals and epidurals) is associated with a lower risk for maternal aspiration and airway compromise, exposes the baby to less anesthetic, and allows for greater maternal involvement in the birth process. For these reasons, it has become the preferred method of anesthesia for cesarean delivery. Spinals that are placed to facilitate cesarean delivery have a duration of one to two hours. Currently, if that duration is exceeded patients must have general endotracheal anesthesia. In addition, suboptimal neuraxial anesthesia for cesarean delivery is not uncommon with an incidence of 2-9%, depending upon the urgency of surgery and the type of neuraxial block. Providing less than adequate anesthesia for cesarean delivery may increase the risk of legal liability. For this reason, some patients with suboptimal neuraxial anesthesia have intraoperative conversion to general endotracheal anesthesia.

The first known description of the use of intraperitoneal local anesthetic to provide anesthesia for cesarean delivery was published in 1975. In this article Ranney et al. described how to use up to 100 mL of 1% procaine to provide anesthesia for cesarean delivery under local field block alone. Some of this was injected into the skin and fascia, and the remainder was diluted to 0.5% and "spilled" into the peritoneum.

Multiple publications have shown that intraperitoneal local anesthetic can be used to treat intraoperative and postoperative pain, prevent postoperative nausea, and shorten hospital length of stay. A recently published 40-month case series showed that chloroprocaine lavage can be used as part of a multimodal approach to treating intraoperative pain. In this case series, the technique of chloroprocaine lavage helped investigators to avoid general endotracheal anesthesia in 32 women having a cesarean delivery.

In this case series, no patients exhibited clinical signs of systemic local anesthetic toxicity. It is believed that chloroprocaine has a limited potential for toxicity because of its short plasma half-life, which is only 11-21 seconds. The purpose of this study is to determine the amount of chloroprocaine that is taken up into the blood stream after intraperitoneal administration to ensure that blood levels are low and do not raise a safety concern. Data obtained from this study will help to define a safe dose of chloroprocaine for intraperitoneal administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 to 50 years of age having scheduled cesarean sections on 12C (Labor and Delivery) within Oregon Health & Science University (OHSU).
* Only subjects having spinal anesthesia will be eligible.
* Only subjects that can have a Pfannenstiel incision will be enrolled.

Exclusion Criteria:

* Subjects with chronic narcotic usage
* Subjects that are deemed to need a combined spinal epidural for any reason.
* Subjects who are unable to successfully get a spinal block
* Subjects with known atypical cholinesterase activity
* American Society of Anesthesiologist physical status IV or higher
* Subjects with contraindication to neuraxial anesthesia (coagulopathy, infection)
* Subjects with stage 4 chronic kidney disease or worse (eGFR < 30 ml/min)
* Subjects with significant hepatic dysfunction (AST or ALT > 2x the upper limit of normal)
* Subjects with allergies to drugs required for this protocol.
* Subjects with multifetal gestations
* Subjects with a BMI > 40 kg/m2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Togioka, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU Labor and Delivery; Oregon Health and Science University Hospital, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranney B, Stanage WF. Advantages of local anesthesia for cesarean section. Obstet Gynecol. 1975 Feb;45(2):163-7. PMID 1118089
- [Derived] Togioka BM, Zarnegarnia Y, Bleyle LA, Koop D, Brookfield K, Yanez ND, Treggiari MM. Pharmacokinetics and Tolerability of Intraperitoneal Chloroprocaine After Fetal Extraction in Women Undergoing Cesarean Delivery. Anesth Analg. 2022 Oct 1;135(4):777-786. doi: 10.1213/ANE.0000000000006064. Epub 2022 May 11. PMID 35544759

RESULTS

PARTICIPANT FLOW:
Groups:
- Preservative Free Chloroprocaine Group 1: 40 ml of preservative-free 1% chloroprocaine administered into the peritoneal cavity after delivery of the baby
- Preservative Free Chloroprocaine Group 2: 40 ml of preservative-free 2% chloroprocaine administered into the peritoneal cavity after delivery of the baby
- Preservative Free Chloroprocaine Group 3: 40 ml of preservative-free 3% chloroprocaine administered into the peritoneal cavity after delivery of the baby
Period: Overall Study
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (6.4) | 34.8 (3.8) | 34 (5.3) | 33.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 15
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 3 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 4 | 4 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15
American Society of Anesthesiologists Physical Status [Count of Participants; unit: Participants] — American Society of Anesthesiologist Physical Status 1 (healthiest/lowest risk patient): A normal healthy patient with no acute or chronic diseases.
  American Society of Anesthesiologist Physical Status 2 (middle risk patient): A patient with mild systemic disease that does not cause functional limitations.
  American Society of Anesthesiologist Physical Status 3 (least healthy/highest risk patient in the study): A patient with severe systemic disease that causes substantial functional limitations
  Participants
    American Society of Anesthesiologists Physical Status 2 | 4 | 4 | 4 | 12
    American Society of Anesthesiologists Physical Status 3 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Chloroprocaine Plasma Concentration at 1 Minute
Description: The chloroprocaine plasma concentration obtained from a venous sample 1 minute after intraperitoneal chloroprocaine administration.
Time Frame: 1 minute after intraperitoneal chloroprocaine administration
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
ng/ml | 14.3 [0.4 to 39.9] | 7.5 [1.0 to 16.6] | 3.5 [1.1 to 6.0]

2. Primary Outcome: Chloroprocaine Plasma Concentration at 5 Minutes
Description: The chloroprocaine plasma concentration obtained from a venous sample 5 minutes after intraperitoneal chloroprocaine administration.
Time Frame: 5 minutes after intraperitoneal chloroprocaine administration
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
ng/ml | 14.5 [4.1 to 24.7] | 14.1 [4.7 to 24.0] | 323.1 [34.8 to 611.4]

3. Primary Outcome: Chloroprocaine Plasma Concentration at 10 Minutes
Description: The chloroprocaine plasma concentration obtained from a venous sample 10 minutes after intraperitoneal chloroprocaine administration.
Time Frame: 10 minutes after intraperitoneal chloroprocaine administration
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
ng/ml | 10.4 [5.8 to 15.1] | 6.0 [1.1 to 10.8] | 217.9 [11.0 to 606.3]

4. Primary Outcome: Chloroprocaine Plasma Concentration at 20 Minutes
Description: The chloroprocaine plasma concentration obtained from a venous sample 20 minutes after intraperitoneal chloroprocaine administration.
Time Frame: 20 minutes after intraperitoneal chloroprocaine administration
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
ng/ml | 2.2 [0.5 to 4.4] | 1.7 [1.0 to 2.7] | 3.4 [0.7 to 7.8]

5. Primary Outcome: Chloroprocaine Plasma Concentration at 30 Minutes
Description: The chloroprocaine plasma concentration obtained from a venous sample 30 minutes after intraperitoneal chloroprocaine administration.
Time Frame: 30 minutes after intraperitoneal chloroprocaine administration
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
ng/ml | 3.4 [0.2 to 9.1] | 1.2 [0.5 to 2.3] | 3.1 [0.6 to 5.5]

6. Other Pre Specified Outcome: Dizziness
Description: description of dizziness upon research coordinator query
Time Frame: Within 4 hours of intraperitoneal chloroprocaine administration
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
Participants | 1 | 0 | 0

7. Other Pre Specified Outcome: Metallic Taste
Description: description of metallic taste upon research coordinator query
Time Frame: within 4 hours of study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
Participants | 0 | 1 | 0

8. Other Pre Specified Outcome: Nausea
Description: description of nausea upon research coordinator query
Time Frame: Within 4 hours of study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
Number analyzed (Participants) | 5 | 5 | 5
Participants | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Preservative Free Chloroprocaine Group 1 | Preservative Free Chloroprocaine Group 2 | Preservative Free Chloroprocaine Group 3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 1/5 | 2/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preservative Free Chloroprocaine Group 1 (N=5) | Preservative Free Chloroprocaine Group 2 (N=5) | Preservative Free Chloroprocaine Group 3 (N=5)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
metallic taste (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03760718/Prot_SAP_000.pdf